CLINICAL TRIAL: NCT00844545
Title: An Open-Label, Multi-Center Controlled Clinical Trial of Eculizumab in Adult Patients With Plasma Therapy-Resistant Atypical Hemolytic Uremic Syndrome (aHUS)
Brief Title: Open Label Controlled Trial of Eculizumab in Adult Patients With Plasma Therapy-Resistant aHUS
Acronym: aHUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C08-002A; BB-IND-11075; EudraCT Number 2008-006952-23
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-06

CONDITIONS: Atypical Hemolytic Uremic Syndrome
Keywords: aHUS
MeSH Terms: conditions — Atypical Hemolytic Uremic Syndrome | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — All patients received open-label eculizumab administered intravenously on the following dose schedule: Induction dose - 900 mg per week for four weeks and a dose of 1200 mg one week later; Maintenance dose - 1200 mg every two weeks. Patients who received plasma exchange or infusion during the eculizumab treatment period received a supplemental dose of 600 mg within one hour before plasma infusion or within one hour after the completion of each plasma exchange

SUMMARY:
The purpose of this study is to determine whether eculizumab is safe and effective in the treatment of adult patients with plasma therapy-resistant Atypical Hemolytic-Uremic Syndrome (aHUS).

ELIGIBILITY:
Exclusion Criteria:

1. TTP, (defined as ADAMTS-13 activity <5%) from an historical observation (prior to initiation of plasma therapy) or as tested at the screening visit by the central laboratory
2. Malignancy within 5 years of screening
3. Typical HUS (Shiga toxin +)
4. Known HIV infection
5. Identified drug exposure-related HUS.
6. Infection-related HUS
7. HUS related to bone marrow transplant
8. HUS related to vitamin B12 deficiency
9. Renal function status requiring chronic dialysis
10. Patients with a confirmed diagnosis of sepsis
11. Presence or suspicion of active and untreated systemic bacterial infection that, in the opinion of the Investigator confounds an accurate diagnosis of aHUS or impedes the ability to manage the aHUS disease
12. Pregnancy or lactation
13. Unresolved meningococcal disease
14. Known Systemic Lupus Erythematosus (SLE) or antiphospholipid antibody positivity or syndrome
15. Any medical or psychological condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study
16. Patients who have received previous treatment with eculizumab
17. Patients receiving IVIG within 8 weeks or Rituximab therapy within 12 weeks of screening.
18. Patients receiving other immunosuppressive therapies such as steroids, mTOR inhibitors or tacrolimus are excluded unless: [1] part of an established post-transplant anti-rejection regime, [2] patient has confirmed anti-CFH antibody requiring immunosuppressive therapy, and [3] dose of such medications have been unchanged for at least 4 weeks prior to the screening period or [4] patient is experiencing an acute aHUS relapse immediately after transplant
19. Patients receiving Erythrocyte Stimulating Agents (ESAs) unless already on a stable dose for at least 4 weeks prior to the screening period, or a washout period of at least 2 weeks from the last dose of ESA therapy.
20. Participation in any other investigational drug trial or exposure to other investigational agent, device, or procedures beginning 4 weeks prior to screening and throughout the entire trial.
21. Hypersensitivity to eculizumab, to murine proteins or to one of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - Atlanta, Georgia
  - Fort Wayne, Indiana
  - New York, New York
  - Grapevine, Texas
  - Houston, Texas
- Innsbruck, Austria
- France (7):
  - Bordeaux
  - Lyon
  - Nantes
  - Paris
  - Quimper
  - Saint-Priest-en-Jarez
  - Tours
- Germany (2):
  - Aachen
  - Essen
- Newcastle, United Kingdom

REFERENCES:
- [Derived] Pugh D, O'Sullivan ED, Duthie FA, Masson P, Kavanagh D. Interventions for atypical haemolytic uraemic syndrome. Cochrane Database Syst Rev. 2021 Mar 23;3(3):CD012862. doi: 10.1002/14651858.CD012862.pub2. PMID 33783815
- [Derived] Legendre CM, Licht C, Muus P, Greenbaum LA, Babu S, Bedrosian C, Bingham C, Cohen DJ, Delmas Y, Douglas K, Eitner F, Feldkamp T, Fouque D, Furman RR, Gaber O, Herthelius M, Hourmant M, Karpman D, Lebranchu Y, Mariat C, Menne J, Moulin B, Nurnberger J, Ogawa M, Remuzzi G, Richard T, Sberro-Soussan R, Severino B, Sheerin NS, Trivelli A, Zimmerhackl LB, Goodship T, Loirat C. Terminal complement inhibitor eculizumab in atypical hemolytic-uremic syndrome. N Engl J Med. 2013 Jun 6;368(23):2169-81. doi: 10.1056/NEJMoa1208981. PMID 23738544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: C08-002A/B combined 2 studies: one for adults (C08-002A, N=16) and one for adolescents (C08-002B, N=1) Please refer to NCT00844844 for combined studies with enrollment number corresponding to each individual study
Pre-assignment Details: Patients had to exhibit a decrease in platelet count despite at least 4 Plasma Therapy (PT) treatments in the 1 week immediately prior to screening. Patients who met the eligibility criteria during screening were enrolled into the Treatment Period which commenced with the first eculizumab dose.
Period: Screening Period
Arm/Group | Eculizumab
Started | 17
Completed | 17
Not Completed | 0
Period: Treatment Period (26 Weeks)
Arm/Group | Eculizumab
Started | 17
Completed | 15
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Period: Extension Treatment Period
Arm/Group | Eculizumab
Started | 13
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 2
Period: Post Treatment Period
Arm/Group | Eculizumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all patients who received any amount of eculizumab, and were considered evaluable for safety and efficacy analyses. For both the efficacy and safety analyses, all 17 patients who were treated with study drug were included in the ITT population.
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet Count Change From Baseline to 26 Weeks
Time Frame: From Baseline to 26 weeks
Population: Change from baseline platelet counts were analyzed for the ITT population using a repeated measurement ANOVA model. A least squares (LS) mean for the change from baseline was produced for each study day for which a measurement of platelet count was scheduled. Significance of change was assessed at the 5% level at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
10^9 cells/L | 65.18 [37.01 to 93.36]
Statistical Analysis 1: Comparison: Eculizumab; With at least 12 patients enrolled and assuming a null hypothesis of no post-dose change from baseline in mean platelet count, the study had approximately 88% power to detect as statistically significant an effect size (mean change from baseline/standard deviation) of at least 1 when using a one sample t-test with a two-sided α=0.05. All analyses were based on the pooled data from the two protocols: C08-002A (adult) and C08-002B (adolescent), a similar protocol, for patients <18 years with aHUS; Test type: Superiority or Other; p < 0.0001, ANOVA; Change from baseline were analyzed using a repeated measurement ANOVA model with time and baseline as fixed effects and subject as a random effect; LS mean change from baseline = 65.18, 95% CI 2-sided [37.01 to 93.36]

2. Primary Outcome: Percentage of Patients With Platelet Count Normalization
Description: The primary objective of the study (per protocol) was to assess the effect of eculizumab to reduce TMA as measured by platelet count change from baseline (BL) during the Treatment Period (26 weeks) in patients with plasma therapy (PT)-resistant aHUS (protocol defined), including assessment of the proportion of patients who achieved Platelet Count Normalization from baseline through 26 weeks. Platelet Count Normalization was defined as the platelet count observed to be ≥150 x 10^9/L on at least two consecutive measurements which span a period of at least four weeks.
Time Frame: Through 26 weeks
Population: The Tabulations of the proportion of patients who achieved platelet count normalization through 26 weeks were performed for the ITT population. Exact binomial confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Percentage of Participants | 82 [57 to 96]
Statistical Analysis 1: Comparison: Eculizumab; All analyses were based on the pooled data from the two protocols: protocol C08-002A for adult patients with aHUS and protocol C08-002B, a similar protocol, for patients < 18 years of age for adolescent patients with aHUS; Test type: Superiority or Other; Percent of platelet count normalization = 82, 95% CI 2-sided [57 to 96]

3. Primary Outcome: Percentage of Patients With Hematologic Normalization
Description: Hematologic Normalization was defined as normalization of both platelet count and lactic dehydrogenase (LDH) sustained for at least two consecutive measurements which spanned a period of at least four weeks.
Time Frame: Through 26 weeks
Population: Tabulations of the proportion of patients who achieved a hematologic normalization through 26 weeks were performed for the ITT population. Exact binomial confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Percentage of Participants | 76 [50 to 93]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of hematologic normalization = 76, 95% CI 2-sided [50 to 93]

4. Secondary Outcome: Percentage of Patients With Complete TMA Response
Description: The proportion of patients who achieved a Complete TMA Response from baseline through 26 weeks of treatment with eculizumab was determined. Complete TMA Response was defined as Hematologic Normalization plus improvement in renal function (defined as as ≥25% reduction from baseline in serum creatinine), which was sustained for two consecutive measurements over a period of at least four weeks.
Time Frame: Through 26 weeks
Population: Tabulations of the proportion of patients who achieved a complete TMA response from baseline through 26 weeks were performed. For this endpoint, for any relevant proportions, exact binomial confidence intervals were produced.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Percentage of Participants | 65 [38 to 86]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of complete TMA response = 65, 95% CI 2-sided [38 to 86]

5. Secondary Outcome: TMA Intervention Rate
Description: TMA Intervention Rate (# PE/PI and # Dialysis Events/Patient/Day) in the eculizumab treatment period (from baseline through 26 weeks) for PE/PI and (from the fifteenth day following the first eculizumab dose through 26 weeks) for new dialysis events was compared with the TMA Intervention Rate during the pre-eculizumab treatment period.
Time Frame: Through 26 weeks
Population: A signed rank test assessed differences in magnitudes of change in TMA intervention rate between the pre-eculizumab treatment period and during eculizumab treatment period for ITT population.
Measure: Mean (Standard Deviation); unit: # events/patient/day
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
# events/patient/day | 0.04 (0.10)
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.78

6. Secondary Outcome: Platelet Count Change From Baseline to 156 Weeks
Time Frame: From Baseline to 156 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: 10^9 cells/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
10^9 cells/L | 111.62 [98.12 to 125.13]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; LS mean change from baseline = 111.62, 95% CI 2-sided [98.12 to 125.13]

7. Secondary Outcome: Percentage of Patients With Platelet Count Normalization
Description: Platelet Count Normalization was defined as the platelet count observed to be ≥150 x 10^9/L on at least two consecutive measurements which span a period of at least four weeks.
Time Frame: Through End of Study, Median Exposure 100.29 Weeks
Population: The Tabulations of the proportion of patients who achieved platelet count normalization through end of the study were performed for the ITT population. Exact binomial confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Percentage of Participants | 88 [64 to 99]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of platelet count normalization = 88, 95% CI 2-sided [64 to 99]

8. Secondary Outcome: Percentage of Patients With Hematologic Normalization
Description: as for outcome 3
Time Frame: Through End of Study, Median Exposure 100.29 Weeks
Population: Tabulations of the proportion of patients who achieved a hematologic normalization through end of study were performed for the ITT population. Exact binomial confidence intervals were produced for the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Percentage of Participants | 88 [64 to 99]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of hematologic normalization = 88, 95% CI 2-sided [64 to 99]

9. Secondary Outcome: Percentage of Patients With Complete TMA Response
Description: The proportion of patients who achieved a Complete TMA Response from baseline through end of the study was determined. Complete TMA Response was defined as Hematologic Normalization plus improvement in renal function (defined as ≥25% reduction from baseline in serum creatinine), which was sustained for two consecutive measurements over a period of at least four weeks.
Time Frame: Through End of Study, Median Exposure 100.29 Weeks
Population: Tabulations of the proportion of patients who achieved a complete TMA response from baseline through end of study were performed. For this endpoint, for any relevant proportions, exact binomial confidence intervals were produced.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
Percentage of Participants | 76 [50 to 93]
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Percent of complete TMA response = 76, 95% CI 2-sided [50 to 93]

10. Secondary Outcome: TMA Intervention Rate
Description: TMA Intervention Rate (# PE/PI and # Dialysis Events/Patient/Day) in the eculizumab treatment period (from baseline through end of the study) for PE/PI and (from the fifteenth day following the first eculizumab dose through end of the study) for new dialysis events was compared with the TMA Intervention Rate during the pre-eculizumab treatment period.
Time Frame: Through End of Study, Median Exposure 100.29 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: # events/patient/day
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
# events/patient/day | 0.04 (0.11)
Statistical Analysis 1: Comparison: Eculizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.78

11. Secondary Outcome: Pharmacokinetics (PK) and Pharmacodynamics (PD); Minimum and Maximum Blood Concentration
Time Frame: Induction Phase for 4 weeks followed by Maintenance Phase starting on Week 5 through 26 weeks or longer.
Population: PK parameters Cmin and Cmax were estimated using a population PK model developed from the observed PK concentration data
Measure: Mean (Standard Deviation); unit: micrograms/mil
Arm/Group | Eculizumab
Number analyzed (Participants) | 17
micrograms/mil
  max concentration during induction period | 145.16 (26.56)
  min concentration during induction period | 93.66 (22.10)
  max concentration during maintenace | 345.14 (89.74)
  Min concentration during maintenance | 151.80 (68.16)

ADVERSE EVENTS:
Time Frame: Through end of study; Exposure to eculizumab in this study extended for a median of 100 weeks and ranged from two weeks to 186 weeks.
Description: At every visit, patients were asked a standard non-leading question to elicit any changes in their medical well-being including inquiry about any hospitalization, accidents, and new or changed concomitant medication regimens. AEs were also documented from any data collected (e.g. laboratory values, physical examination findings, ECG changes, etc.).
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 17/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Transplant rejection (Immune system disorders) | 1
asymptomatic bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 3
Adenomyosis (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Dysponea (Respiratory, thoracic and mediastinal disorders) | 1
Accelerated hypertension (Vascular disorders) | 2
Embolism venous (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Malignant hypertension (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cushingold (Endocrine disorders) | 1
Hyperparathyroidism secondary (Endocrine disorders) | 1
Hypothalamo-pituitary disorder (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 8
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oral pain (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Cyst (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 3
Influenza like illness (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 3
Pyrexia (General disorders) | 3
Tenderness (General disorders) | 1
Thirst (General disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Camylobacter infection (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Genital herpes (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Onychomycosis (Infections and infestations) | 1
Papilloma viral infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Urinary tract infection bacterial (Infections and infestations) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Eye injury (Injury, poisoning and procedural complications) | 1
Incision site oedema (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 2
Muscle rupture (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Antibiotic resistant Staphylococcus test positive (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Carbon dioxide abnormal (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Haptoglobin decreased (Investigations) | 1
Reticulocyte count increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Iron deficiency (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sinus headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Dysthymic disorder (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Renal pain (Renal and urinary disorders) | 1
Adenomyosis (Reproductive system and breast disorders) | 1
Breast calcifications (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Metrorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 2
Uterine malposition (Reproductive system and breast disorders) | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Skin depigmentation (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Tooth extraction (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
Poor venous access (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in this multicenter study involved a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis.